CLINICAL TRIAL: NCT05481463
Title: A Open-label, Single-arm, Single-center, Phase II Clinical Study of Surufatinib Combined With TAS-102 in Third-line and Later-line Therapy of Patients With Advanced Pancreatic Cancer
Brief Title: Surufatinib Combined With TAS-102 in Third-line and Later-line Therapy of Patients With Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Dong sheng Zhang, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SPRING-P104
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-03

CONDITIONS: Pancreatic Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — surufatinib; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- surufatinib combined with TAS-102 (Experimental): Surufatinib 250mg,TAS-102 35mg/m2
  Interventions: Drug: Surufatinib; Drug: TAS-102

INTERVENTIONS:
Drug: Surufatinib — surufatinib,250mg, qd, po, 28 days for a cycle
Drug: TAS-102 — TAS-102,35mg/m2, po, d1-5, d8-12, bid, 28 days for a cycle

SUMMARY:
This is a single-center, single-arm, open-label, phase 2 clinical study, to explore the efficacy and safety of surufatinib combined with TAS-102 in third-line and later-line therapy of patients with advanced pancreatic cancer

DETAILED DESCRIPTION:
surufatinib:250mg,QD,Q4W TAS-102:35mg/m2,D1-5,D8-12,Q4W

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent has been signed
2. Histologically or cytologically confirmed unresectable, locally advanced or metastatic pancreatic cancer
3. Age ≥ 18 years, ≤75 years, male or female
4. ECOG PS：0-1, expected overall survival ≥12 months
5. Patients who have previously received at least two systemic therapies for locally advanced or metastatic pancreatic cancer; patients with BRCA1/2 germline mutations have previously received platinum-containing regimens
6. Patients must have at least one measurable liver metastases (RECIST 1.1)
7. No serious organic diseases of the heart, lungs, brain and other organs
8. Patients must have adequate organ and bone marrow function
9. Women of childbearing age must have a negative pregnancy test within the first day of the study, and contraceptive methods should be taken during the study until 6 months after the last administration

Exclusion Criteria:

1. Participated in clinical trials of other anti-tumor drugs within 4 weeks before enrollment
2. Previously received VEGFR inhibitors or immune checkpoint inhibitors
3. Patients had other malignant tumors in the past 5 years, except for the cured skin basal cell carcinoma and cervical carcinoma in situ
4. Patients previously had brain metastasis or current brain metastasis
5. Received any operation (except biopsy) or invasive treatment or operation (except venous catheterization, puncture and drainage, internal/external drainage surgery for obstructive jaundice, etc.) within 4 weeks before enrollment
6. Clinically significant electrolyte abnormality
7. Patient currently has uncontrolled hypertension, defined as: systolic blood pressure > 140mmHg or diastolic blood pressure > 90mmHg
8. Proteinuria ≥ 2+ (1.0g/24hr)
9. Patients whose tumor is highly likely to invade important blood vessels and cause fatal hemorrhage during the follow-up study as judged by the investigator
10. Have evidence or history of bleeding tendency within 3 months, significant bleeding symptoms or a clear bleeding tendency within 3 months before enrollment
11. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within 6 months before enrollment; NYHA classification > 2 Grade; ventricular arrhythmia requiring medical therapy; ECG showing QTc interval ≥ 480 ms
12. Active or uncontrolled serious infection (≥CTCAE grade 2 infection)
13. Unrelieved toxic reactions ≥ CTCAE grade 2 due to any previous anticancer treatment, excluding alopecia, lymphopenia and neurotoxicity of ≤ grade 2 caused by oxaliplatin
14. Pregnant or lactating women
15. Any other disease, with clinically significant metabolic abnormalities, physical examination abnormalities or laboratory abnormalities, according to the judgment of investigator that the patient is not suitable for the the study drug (such as having epileptic seizures and require treatment), or would affect the interpretation of study results, or put patients at high risk
16. Clinical confirmed human immunodeficiency virus (HIV) infection, history of clinically significant liver disease, including viral hepatitis (hepatitis B / C (HBV DNA Positive[1×104 copies/mL or >2000 IU/ml], HCV RNA positive[>1×103 copies/mL]), or other hepatitis, cirrhosis])
17. Patients with autoimmune disease or suspected autoimmune disease (including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, enteritis, multiple Sclerosis, vasculitis, glomerulonephritis, uveitis, hypophysitis, hyperthyroidism, etc.)
18. Patients who are allergic or suspected to be allergic to the study drug or similar drugs
19. Patients have other factors that may affect the results of the study or cause the study to be terminated halfway, such as alcoholism, drug abuse, other serious diseases (including mental diseases) that require concomitant treatment, and serious laboratory abnormalities. Accompanied by family or social factors, which will affect the safety of patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-05-10 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | up to 24 months
  PFS is defined as the time from enrollment to the first documented disease progression or death due to any cause, whichever occurs first. Responses are according to the Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by investigator

SECONDARY OUTCOMES:
disease control rate (DCR) | up to 24 months
  DCR was defined as the percentage of participants who have a confirmed complete response（CR） or partial response（PR） or stable disease（SD） per RECIST 1.1 as assessed by investigator
overall survival (OS) | up to 24 months
  OS is the time from enrollment to death due to any cause.
objective response rate (ORR) | up to 24 months
  Defined as percentage of participants achieving assessed complete response (CR) and partial response (PR) by the investigator according to the RECIST 1.1.
quality of life (QoL) | up to 24 months
  Assessing the quality of life of cancer patients by QLQ-C30
adverse events (AE) | up to 24 months
  overall incidence of adverse events (AE); incidence of grade 3 or higher AE; incidence of severe adverse events (SAE); incidence of AEs leading to discontinuation of drug use; incidence of AEs leading to suspension of drug use.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Zhang, PhD, Principal Investigator — Sun Yat-sen University Cancer Center, State Key Laboratory of Oncology in South China
Locations (1):
- Cancer center of SunYat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lu Y, Lin Q, Mo Y, Liu F, Zhang M, Huang R, Wang Y, Wang Y, Wang Z, Luo H, Guo G, Chen J, Liu Y, He M, Wang F, Wang F, Zhang D. Efficacy and safety of TAS-102 plus Surufatinib in third and later line metastatic pancreatic cancer: a prospective, single center and biomarker exploratory, phase II study. Mol Cancer. 2025 Oct 2;24(1):235. doi: 10.1186/s12943-025-02437-0. PMID 41039600